CLINICAL TRIAL: NCT01273168
Title: Phase I Trial of Z-Endoxifen in Adults With Refractory Hormone Receptor-Positive Breast Cancer, Desmoid Tumors, Gynecologic Tumors, or Other Hormone Receptor-Positive Solid Tumors
Brief Title: Endoxifen in Adults With Hormone Receptor Positive Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110061; 11-C-0061
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hormone Receptor-Positive Breast; Gynecologic; Desmoid; Hormone Receptor-Positive Neoplasms
Keywords: Pharmacokinetics; Advanced Cancer; Cytochrome P450; Selective Estrogen Receptor Modulator; Tamoxifen Metabolite; Gynecologic Cancer; Breast Cancer; Desmoid Tumor; Endometrial Cancer; Ovarian Cancer; Uterine Cancer; Fallopian Tube Cancer; Peritoneal Cancer
MeSH Terms: conditions — Desmoid Tumors; Breast Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Uterine Neoplasms; Fallopian Tube Neoplasms | interventions — 4-hydroxy-N-desmethyltamoxifen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Z-endoxifen will be administered orally once a day in 28-day cycles
  Interventions: Drug: Z-Endoxifen

INTERVENTIONS:
Drug: Z-Endoxifen — Genetic polymorphisms in CYP2D6 and concomitant medications alter tamoxifen metabolism, limiting exposure to the active metabolite endoxifen. These factors are associated with a higher rate of recurrence and shorter disease-free survival in breast cancer patients receiving tamoxifen. Administration of endoxifen directly to patients is anticipated to bypass the effects of CYP2D6 polymorphisms and concomitant medications and provide adequate active drug levels in all treated patients, resulting in clinical benefit.

SUMMARY:
Background:

* Some types of cancer cells that have hormone receptors on their surfaces need the hormone estrogen to grow. The drug tamoxifen blocks estrogen from binding to the tumor cells, which helps to slow or stop the growth of cancer. Tamoxifen has been approved for treatment of certain types of estrogen-linked cancers, such as breast and ovarian cancer.
* The experimental drug Z-Endoxifen HCl (endoxifen) is related to tamoxifen, and has been shown to work against similar estrogen-linked cancers. In many cancer patients, tamoxifen is turned into endoxifen by enzymes in the liver; however, not all people have the liver enzymes that can turn tamoxifen into endoxifen, which means that the drug cannot work properly. Taking certain other drugs at the same time as tamoxifen can also keep it from turning into endoxifen. Researchers are interested in determining whether endoxifen tablets are effective in slowing or stopping tumor growth in individuals whose hormone-linked tumors have not responded to standard treatment.

Objectives:

- To test the safety and effectiveness of daily endoxifen in individuals with hormone receptor positive solid tumors that have not responded to standard treatment.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with hormone receptor positive solid tumors (breast or other tumors), desmoid tumors, or gynecologic tumors that have not responded to standard treatment.

Individuals with breast cancer must have had at least one prior chemotherapy regimen and one prior hormonal regimen for metastatic disease.

Design:

* Participants will be screened with a full medical history (including prior hormone use) and physical examination, as well as blood and urine tests, tumor imaging studies, and an eye examination.
* Participants will take endoxifen tablets daily for 28-day cycles of treatment, and will be asked to keep a medication diary to record any side effects.
* Participants will have regular clinic visits with blood and urine samples and imaging studies to evaluate the cancer's response to treatment.
* Participants will continue to take endoxifen for as long as the cancer responds to the treatment.

DETAILED DESCRIPTION:
Background:

Genetic polymorphisms in CYP2D6 and concomitant medications alter tamoxifen metabolism, limiting exposure to the active metabolite endoxifen. These factors are associated with a higher rate of recurrence and shorter disease-free survival in breast cancer patients receiving tamoxifen.

Administration of endoxifen directly to patients is anticipated to bypass the effects of CYP2D6 polymorphisms and concomitant medications and provide adequate active drug levels in all treated patients, resulting in clinical benefit.

16 alpha-[18F]-fluoro-17 beta-estradiol (FES) is an investigational radiolabeled imaging agent used with positron emission tomography (PET) to investigate tumor estrogen receptor activity.

Objectives:

Primary:

Establish the safety and tolerability of oral endoxifen (Z-Endoxifen HCl) administered on a daily schedule to patients with refractory hormone receptor-positive solid tumors (breast or other tumors), desmoid tumors, or gynecologic tumors.

Establish the maximum tolerated dose (MTD) of oral Z-endoxifen HCl administered on a daily schedule.

Secondary:

Determine the pharmacokinetics of oral Z-endoxifen (HCl form).

Exploratory:

Evaluate the change in [18F]FES uptake using PET/CT in hormone receptor-positive tumors before and after treatment with oral Z endoxifen HCl.

Eligibility:

Adults with histologically documented hormone receptor-positive solid tumors (breast or other tumors), desmoid tumors, or gynecologic tumors.

Patients with breast cancer must have had at least one prior chemotherapy regimen and one prior hormonal regimen for metastatic disease. All other patients must have disease that has progressed following at least one line of standard therapy.

No major surgery, radiation, hormonal, or chemotherapy within 4 weeks prior to study enrollment, and recovered from toxicities of prior therapies to at least eligibility levels.

Patients in the 6-patient expansion cohort at the MTD will be asked to undergo optional tumor biopsies for research purposes.

Study Design:

Z-endoxifen will be administered orally once a day in 28-day cycles.

Dose escalation will proceed until the MTD is established or targeted maximum dose (DL8) reached. Six additional patients will then be entered in an expansion cohort to assess pharmacodynamics and pharmacokinetics.

When imaging agent is available, optional FES PET/CT scans will be performed at baseline and 1-3 hours after Z-endoxifen treatment once during week 1 of cycle 1.

As a relative bioavailability study, 6 patients in the expansion cohort will be given a single dose of the free base form of Z-endoxifen on day 1 and will then continue on study taking Z-endoxifen HCl; blood and urine will be collected for PK at baseline, on cycle 1 days 1 and 2, and on cycle 2 day 1. Please note: As of Febuary 2017, we will no longer evaluate the free base form of Z-endoxifen in the expansion cohort due to drug supply issues.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with the following types of histologically documented solid tumors:

* ER +/PR+, ER+/PR-, or ER-/PR+ breast cancer
* Gynecologic tumors (endometrial, ovarian, uterine, fallopian tube, peritoneal, etc.)
* Desmoid tumors
* Tumors that are ER+ or PR+ by immunohistochemistry (including low-level expression) such as non-small cell lung, colorectal, and prostate

Patients with breast cancer must have had at least one prior chemotherapy regimen for metastatic disease. Additionally, patients with breast cancer must have received prior tamoxifen and/or aromatase inhibitor therapy (if postmenopausal) with at least one hormonal regimen in the metastatic setting. Patients with HER2+ breast cancer must have progressed after at least one prior HER2-directed regimen (trastuzumab, lapatinib) for metastatic disease.

All other patients must have disease that has progressed following at least one line of standard therapy. Prior therapy with tamoxifen is allowed.

Patients enrolled based on tumor ER/PR status must have ER/PR status confirmed by the Laboratory of Pathology, NIH. ER/PR status will be determined on a metastatic site, if possible; otherwise, the original site or available tissue will be acceptable.

Patients must have recovered to at least eligibility levels following any display of adverse events and/or toxicity due to prior chemotherapy or biologic therapy. They must not have had hormonal therapy, chemotherapy or biologic therapy within 4 weeks prior to entering the study (6 weeks for nitrosoureas or mitomycin C, or UCN-01). Patients must be greater than or equal 2 weeks since any prior administration of study drug in a Phase 0 study (also referred to as an "early Phase I study" or "pre-Phase I study" where a sub-therapeutic dose of drug is administered) at the PI's discretion. Patients must be greater than or equal to 4 weeks since any prior radiation or major surgery. However, patients receiving bisphosphonates or therapeutic anticoagulation are eligible for this trial.

Age greater than or equal 18 years

The Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2

Life expectancy > 3 months

Patients must have normal or adequate organ and marrow function as defined below:

Absolute neutrophil count greater than or equal to 1,500/microL

Platelets greater than or equal to 100,000/microL

Total bilirubin within less than or equal to 1.5 times institutional upper limit of normal

AST (SGOT)/ALT (SGPT) less than or equal to 2.5 times institutional upper limit of normal

Creatinine < 1.5 times upper limit of normal

OR

Creatinine clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels greater than or equal to 1.5 times upper limit of normal.

The effects of Z-endoxifen on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate nonhormonal contraception (barrier method of birth control or abstinence) prior to study entry, for the duration of study participation, and for 2 months after discontinuation from the study. Women of childbearing potential must have a negative pregnancy test in order to be eligible. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Z-endoxifen, breastfeeding should be discontinued if the mother is treated with Z-endoxifen.

Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Patients receiving any other investigational agents.

Patients with known brain metastases are excluded from this clinical trial, with the exception of patients whose brain metastatic disease status has remained stable for greater than or equal to 3 months after treatment of the brain metastases, without steroids or anti-seizure medications. These patients may be enrolled at the discretion of the principal investigator.

Patients with clinically significant illnesses which could compromise participation in the study, including, but not limited to, uncontrolled infection, uncontrolled diabetes, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia, stroke/cerebrovascular accident within the past 6 months, or psychiatric illness/social situations that in the investigator s opinion would make it undesirable for the patient to participate in the trial, or which would jeopardize compliance with the protocol.

Patients with untreated spinal cord metastases or metastases close to vital organs (as determined by the principal investigator) are excluded because of the risk of hormonal flare.

Patients with a history of deep vein thrombosis must be on anti-coagulation therapy prior to enrollment. Patients requiring prophylactic anti-coagulation are eligible.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Establish safety and MTD of Z-endoxifen | 28 days (1 cycle)
  Adverse events will be graded as described in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Determine the pharmacokinetics of Z-endoxifen (free base and HCl forms) | 28 days (1 cycle)

CONTACTS AND LOCATIONS:
Overall Officials: Alice P Chen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.@@@@@@All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@Requests for all collected IPD data from clinical trials, conducted under a binding collaborative agreement between NCI/DCTD and a pharmaceutical/biotechnology company, that are not under DSMB monitoring must be in compliance with the terms of the binding collaborative agreement and must be approved by NCI/DCTD and the Pharmaceutical Collaborator.

REFERENCES:
- [Background] Goetz MP, Suman VJ, Reid JM, Northfelt DW, Mahr MA, Ralya AT, Kuffel M, Buhrow SA, Safgren SL, McGovern RM, Black J, Dockter T, Haddad T, Erlichman C, Adjei AA, Visscher D, Chalmers ZR, Frampton G, Kipp BR, Liu MC, Hawse JR, Doroshow JH, Collins JM, Streicher H, Ames MM, Ingle JN. First-in-Human Phase I Study of the Tamoxifen Metabolite Z-Endoxifen in Women With Endocrine-Refractory Metastatic Breast Cancer. J Clin Oncol. 2017 Oct 20;35(30):3391-3400. doi: 10.1200/JCO.2017.73.3246. Epub 2017 Aug 30. PMID 28854070
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0061.html